CLINICAL TRIAL: NCT01226147
Title: Efficacy and Safety of Tamibarotene(AM80) for Lupus Nephritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kinki University (Other)
Responsible Party: Masanori Funauchi, MD, Professor, Department of Nephrology and Rheumatology, Kinki University Faculty of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AM80-F01
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis; SLE; retinoid; tamibarotene
MeSH Terms: conditions — Lupus Nephritis | interventions — tamibarotene

INTERVENTIONS:
Drug: Tamibarotene — 4mg/day for 24 weeks.

SUMMARY:
An open-label study to evaluate the efficacy and safety of orally administered Tamibarotene to patients of Lupus Nephritis

DETAILED DESCRIPTION:
Tamibarotene is a synthetic retinoid presently approved in Japan for the treatment of APL, and in US, Europe and China it is still under development for APL. Compared to other retinoid drugs available, Tamibarotene has not just a higher activity as a retinoid, but also shows a higher receptor selectivity towards the Retinoic Acid Receptor (RAR) subtypes alfa and beta, but not gamma. All trans retinoic acid (ATRA) and its derivatives are usually pan-agonists to these subtypes, and often are know for the irritation to the skin as one of their major side effects which is due to the RAR gamma subtype. Moreover, unlike ATRA tamibarotene does not cause induction of drug metabolism by CRABP.

Tamibarotene is known to moderate T1/T2 balance as well as Treg/Th17 balance through binding RAR-alfa receptor, and shows efficacy to various autoimmune and inflammatory animal models.

In the preliminary clinical research, patients with lupus nephritis for whom prednisolone treatment was not sufficient enough was treated with oral administration of ATRA to show a remarkable decrease in their protein urea (ref. Kinoshita et al, Am.J.Kidney Dis., 2009 Jul 21).

Based on these results, the investigators plan by this study to evaluate the efficacy of tamibarotene together with the safety to the patients of lupus nephritis.

Tamibarotene is used clinically in Japan since 2005. It's side effects are known to be similar to that of other clinically used retinoids.

ELIGIBILITY:
Inclusion Criteria:

* Steroid refractory lupus nephritis

  * more than 10mg of steroid failed to control disease activity
  * patients who failed to reduce the amount of steroid
  * patients who couldn't increase the amount of steroid due to side effects
* Urine Protein creatinine raio > 0.5 or RBC in urine >= 6 /HPF
* Anti dsDNA antibody > 10 IU/ml or complement C3 < 84 mg/dl
* Patients willing to take contraceptive measures throughout the study and for female patients two years after the study and for men six months after the study.

Exclusion Criteria:

* Pregnant or breastfeeding female patients
* Hepatic failure patients
* Triglyceride > 500 mg/dl
* Patients who started the immunosuppressant therapy or increased the amount of immunosuppressant within 8 weeks prior to test drug administration
* Patients who received cyclophosphamide puls within 6 months prior to test drug administration
* Patients with diabetics (HbA1c > 8.0%)
* Serum creatinine ≧1.5mg/dL
* CNS( Central Nerve System) Lupus patients

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Renal Function | 24 weeks
Urinary Protein values | 24 weeks
Urinary Sediment | 28 weeks
Anti di-DNA antibody and complement C3 | 28 weeks

SECONDARY OUTCOMES:
Disease activity index, total improvement | 24 weeks
SLEDAI | 24 weeks
Safety | 28 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kinki University Hospital, Osaka, Japan

REFERENCES:
- [Background] Kinoshita K, Kishimoto K, Shimazu H, Nozaki Y, Sugiyama M, Ikoma S, Funauchi M. Successful treatment with retinoids in patients with lupus nephritis. Am J Kidney Dis. 2010 Feb;55(2):344-7. doi: 10.1053/j.ajkd.2009.06.012. Epub 2009 Jul 23. PMID 19628316